CLINICAL TRIAL: NCT05862298
Title: Pre-Anaesthetic Venous Excess Ultrasound -Score and Their Correlations With the Spinal-Induced Hypotension in Geriatric Patients
Brief Title: Spinal-Induced Hypotension in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Other Study IDs: postspinal hypotension
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Spinal Induced Hypotension; Geriatric Population; Intravascular Volume

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: venous excess ultrasound score — Venous congestion is classified into 4 grades. If the Inferior vena cava is not plethoric, there is deemed to be no congestion (grade 0), and further Doppler examination is not performed. When the IVC is plethoric but there are no severely abnormal waveforms (defined as S-wave reversal on hepatic, >50% pulsatility on portal, and a monophasic pattern on intrarenal Doppler), congestion is considered to be mild (grade 1). Plethoric IVC with at least 1 severely abnormal pattern is considered to be moderate congestion (grade 2), while 2 or more abnormal Doppler patterns constitute severe congestion (grade 3)

SUMMARY:
The study will be conducted to asses preoperative condition of venous system by VExUS score and it's relation with the incidence of spinal induced hypotension in geriatric patients undergoing surgery with spinal anaesthesia.

DETAILED DESCRIPTION:
An assessment of the intravascular volume deficit prior to the spinal anaesthesia conduction may help to predict the occurrence of a critical decrease in blood pressure, so several indices have been proposed to assess it's status depending on either a fluid challenge or an assessment of heart-lung interaction. Heart rate variability, passive leg raise test, and peripheral perfusion index have revealed good abilities to predict spinal induced hypotension. The inferior vena cava (IVC) collapsibility index provides high diagnostic accuracy in predicting spinal induced hypotension The VeXUS score is a four-staged validated protocol which evaluates the presence and severity of systemic venous congestion in the inferior vena cava (IVC) and organs (liver, gut, and kidneys) by evaluating the (IVC) diameter, venous waveforms of the hepatic vein (HV), portal vein (PV), and interlobar renal veins using colour Doppler (CD) and pulsed wave Doppler (PWD)

ELIGIBILITY:
Inclusion Criteria:

* . Patients aging 65 or older
* Lower body surgeries to be done with spinal anaesthesia
* BMI less than 30 kg/m2.
* Patients with ASA I-III

Exclusion Criteria:

* Patient refusal
* Major bloody surgeries (class c surgeries)
* Patients with a history of cardiovascular disorders including arrhythmias, heart failure, tricuspid or mitral regurgitation, dilated right atrium or ventricle, AF
* Patients with a history of respiratory disorders
* Patients with cirrhotic liver
* Patients with pulmonary hypertension
* Patients with renal diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: geriatric patients aged greater 65 years scheduled for Lower body surgeries under spinal anaesthesia with BMI less than 30 kg/m2 with ASA I-III. These populations are high susceptible for development of spinal induced hypotension with high incidence of morbidity and mortality
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
venous excess ultrasound score | immediate preoperative period before the induction of spinal anesthesia
  score used to assess venous circulation

CONTACTS AND LOCATIONS:
Locations (1):
- tarek Abdelhay Mostafa, Tanta, El Gharbyia, Egypt